CLINICAL TRIAL: NCT06511011
Title: Efficacy and Safety of Modified Suan ZaoRen Tang-TianWang BuXin Dan in the Treatment of Chronic Insomnia: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Chinese Medicine in Treating Insomnia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Insomnia study
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mSZT-TBD granules (Experimental): Modified Suan ZaoRen Tang-TianWang BuXin Dan granules
  Interventions: Drug: Modified Suan ZaoRen Tang-TianWang BuXin Dan
- Placebo granules (Placebo Comparator): Placebo granules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modified Suan ZaoRen Tang-TianWang BuXin Dan — Chinese medicine granules for 6 weeks
  Other Names: mSZT-TBD
  Arms: mSZT-TBD granules
Drug: Placebo — Placebo granules for 6 weeks
  Other Names: Placebo granules
  Arms: Placebo granules

SUMMARY:
This is a randomized, double-blinded, placebo-controlled clinical trial. Eligible participants will randomized into either treatment group (CM granules) or placebo group (placebo granules) for 6 weeks, followed by a post-treatment visit at week 9. The primary outcome is the change in Pittsburgh Sleep Quality Index (PSQI) at week 6.

DETAILED DESCRIPTION:
Insomnia is one of the most general health concerns in the society. It is generally defined as a self-reported sleep disorder problem of the patient, characterized by difficulty in falling asleep, or difficulty maintaining sleep. According to American Insomnia Survey, 42.6% of the respondents reported of having at least one of the insomnia symptoms.

Chinese medicine can be an alternative to the treatment of insomnia. Suan Zao Ren Tang and Tian Wang Bu Xin Dan are two of the most common Chinese herbal formulae to treat insomnia, for which Suan Zao Ren Tang has the functions to nourish blood and calm the mind, clear heat and alleviate vexation, and Tian Wang Bu Xin Dan has the function to nourish the heart and calm the mind, and nourish Yin and clear heat. In this study, we will modify the formula of Suan ZaoRen Tang with TianWang BuXin Dan, and observe the effectiveness and safety of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years;
* Eligible for the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, criteria for insomnia disorder. The criteria include having difficulties in falling asleep, difficulties in staying asleep, or early morning awakening with clinically significant consequences for daily life for at least 3 nights per week for at least 6 months;
* Insomnia Severity Index (ISI) total score of at least 8 indicating insomnia at the clinical level;
* Diagnosed to be Yin deficiency-induced internal heat pattern according to traditional Chinese Medicine (TCM) theory;
* Able to complete questionnaires and take medications as scheduled; and
* Voluntary written consent.

Exclusion Criteria:

* Known nervous system disease (eg, stroke, Parkinson's Disease);
* Known mental disorders (eg, depression or anxiety) or HADS score 11 or above in any either item;
* Known sleeping related diseases (eg. sleep apnea, nocturnal myoclonus, restless legs, severe nocturnal enuresis or narcolepsy) that may affect the sleeping quality;
* Known pharmacologically induced insomnia;
* With symptoms that significantly disturb sleep such as pain, fever, diarrhea, frequent micturition, and cough;
* Know treatment to comorbid sleep disorders, such as sleep apnea or narcolepsy;
* Work on shift or on night shift;
* Concomitant pharmacological treatment or herbal medicines for insomnia within the past month;
* Known severe medical conditions, such as cardiovascular, liver, kidney or hematopoietic system disease, diabetes mellitus, cancers, cerebrovascular diseases;
* Impaired hematological profile and liver / renal function exceeds the upper limit of the reference value by 2 times;
* Known alcohol and / or drug abuse;
* Known allergic history to any Chinese herbal medicines;
* Diagnosed to be deficiency of spleen according to TCM theory;
* Any contraindications for taking Chinese medicines in the opinion of the investigators;
* Know pregnant or lactating; and
* Involved in other interventional clinical studies at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The change in Pittsburgh Sleep Quality Index (PSQI) | Week 6
  PSQI, which is a self-reported instrument, is commonly used in assessing the sleep quality in many studies. It consists of 19 items, covering seven domains, including subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
  PSQI items use varying response categories that include recording usual bed time, usual wake time, number of actual hours slept, and number of minutes to fall asleep, as well as forced-choice Likert-type responses (scoring from 1-4, which 1 indicates the best and 4 indicates the worst).

SECONDARY OUTCOMES:
The change in Pittsburgh Sleep Quality Index (PSQI) | Week 3
  PSQI, which is a self-reported instrument, is commonly used in assessing the sleep quality in many studies. It consists of 19 items, covering seven domains, including subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
  PSQI items use varying response categories that include recording usual bed time, usual wake time, number of actual hours slept, and number of minutes to fall asleep, as well as forced-choice Likert-type responses (scoring from 1-4, which 1 indicates the best and 4 indicates the worst).
The change in Pittsburgh Sleep Quality Index (PSQI) | Week 9
  PSQI, which is a self-reported instrument, is commonly used in assessing the sleep quality in many studies. It consists of 19 items, covering seven domains, including subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
  PSQI items use varying response categories that include recording usual bed time, usual wake time, number of actual hours slept, and number of minutes to fall asleep, as well as forced-choice Likert-type responses (scoring from 1-4, which 1 indicates the best and 4 indicates the worst).
Sleep parameter data | From baseline to week 9.
  Wrist actigraphy, which is a small size monitor, is an alternative to objectively measure the sleep patterns of subjects, the measuring parameters include sleep onset latency (SOL), wake time after sleep onset (WASO), total sleep time duration (TST), total time in bed (TIB), and sleep efficiency (SE). The actigraph will be recorded using Philips Actiwatch 2.
The change in Insomnia Severity Index (ISI) | Week 3
  ISI is a self-reported questionnaire to assess both daytime and nighttime components of insomnia. It consists of seven items to evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28
The change in Insomnia Severity Index (ISI) | Week 6
  ISI is a self-reported questionnaire to assess both daytime and nighttime components of insomnia. It consists of seven items to evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28
The change in Insomnia Severity Index (ISI) | Week 9
  ISI is a self-reported questionnaire to assess both daytime and nighttime components of insomnia. It consists of seven items to evaluate the severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28
The change in Hospital Anxiety and Depression Scale (HADS) | Week 3
  HADS consists of 7 depression items and 7 anxiety items which measures the cognitive and emotional aspects of depression and anxiety. The scale is a 4-point Likert scale, ranging from 0 -3. Score range. 0 - 42 for the total score; 0 -21 for the HADS-Anxiety and HADS-Depression.
The change in Hospital Anxiety and Depression Scale (HADS) | Week 6
  HADS consists of 7 depression items and 7 anxiety items which measures the cognitive and emotional aspects of depression and anxiety. The scale is a 4-point Likert scale, ranging from 0 -3. Score range. 0 - 42 for the total score; 0 -21 for the HADS-Anxiety and HADS-Depression.
The change in Hospital Anxiety and Depression Scale (HADS) | Week 9
  HADS consists of 7 depression items and 7 anxiety items which measures the cognitive and emotional aspects of depression and anxiety. The scale is a 4-point Likert scale, ranging from 0 -3. Score range. 0 - 42 for the total score; 0 -21 for the HADS-Anxiety and HADS-Depression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No